CLINICAL TRIAL: NCT01650376
Title: Phase Ib With Expansion of Patients at the MTD Study of Olaparib Plus Weekly (Metronomic) Carboplatin and Paclitaxel in Relapsed Ovarian Cancer Patients
Brief Title: Phase Ib Study of Olaparib Plus Weekly Carboplatin and Paclitaxel in Relapsed Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swedish Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISS22810034
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Uterine Cancer
Keywords: Ovarian Neoplasms; Cancer of the Ovary; Ovarian Cancer; Uterine Neoplasms; Cancer of the Uterus; Uterine Cancer; Olaparib; AZD2281; Carboplatin; Paclitaxel; Relapsed
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms; Recurrence | interventions — olaparib; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib plus carboplatin and paclitaxel (Experimental)
  Interventions: Drug: Olaparib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Olaparib — Olaparib will be administered orally on Days 1, 2, and 3 of each week until DLT or disease progression. A minimum of 3 patients will be enrolled into each cohort. The anticipated dose escalation sequence of olaparib is 50, 100, 150 and 200 mg, taken twice a day will be used.
  Other Names: AZD-2281; AZD2281; AZD 2281
Drug: Carboplatin — AUC 2 weekly for 3 weeks of a 4 week cycle. For patients who experience a complete response, the carboplatin and paclitaxel will be discontinued and olaparib monotherapy (400 mg, taken twice a day) will continue until disease progression and as long as the investigator feels they are benefiting from the treatment.
  Other Names: Paraplatin; Paraplatin NovaPlus
Drug: Paclitaxel — 60mg/m2 weekly for 3 weeks of a 4 week cycle. For patients who experience a complete response, the carboplatin and paclitaxel will be discontinued and olaparib monotherapy (400 mg, taken twice a day) will continue until disease progression and as long as the investigator feels they are benefiting from the treatment.
  Other Names: Taxol; Onxol; Nov-Onxol; Paclitaxel Novaplus

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of the investigational agent, olaparib, to give in combination with carboplatin and paclitaxel in patients with relapsed ovarian cancer or uterine cancer. Furthermore, the investigators intend to study the safety and tolerability of the study treatment, response to treatment, time to disease progression, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (stage III or IV), histologically or cytologically documented ovarian cancer or serious uterine cancer patients who relapsed after primary therapy with a platinum and a taxane. This includes:

  * Platinum sensitive: relapsed at least 6 months following platinum treatment
  * Platinum refractory: the cancer grew while on platinum treatment
  * Platinum resistant: recurrence within 6 months of platinum treatment
* Must have failed first line treatment
* ECOG performance status 0-2
* Must be able to swallow and retain oral medication
* Life expectancy greater than 16 weeks
* Must have normal organ and bone marrow function defined as follows:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * White blood cells (WBC) > 3 x 10^9/L
  * Platelet count ≥ 100 10^9/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5 ULN
  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)

Exclusion Criteria:

* Any previous treatment with a PARP inhibitor, including olaparib
* Any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or longer period depending on the defined characteristics of the agents used)
* Currently receiving the following classes of inhibitors of CYP3A4: azole antifungals, macrolide antibiotics, and protease inhibitors
* Second primary cancer except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* Symptomatic uncontrolled brain metastases
* Major surgery within 2 weeks of starting study treatment
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Known active hepatic disease (i.e. Hepatitis B or C)
* Uncontrolled seizures
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin or paclitaxel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | 1 cycle (1 cycle = 28 days)

SECONDARY OUTCOMES:
Number of Reported Adverse Events | Weekly assessments of clinical and laboratory values, and vital sign measurements performed while receiving study treatment. (Anticipated time of 6 months)

OTHER OUTCOMES:
Response to Therapy | Measured by CT scans performed every 8 weeks while receiving treatment. (Anticipated time of 6 months)
Time to Progression | Measured by CT scans performed every 8 weeks while receiving treatment. (Anticipated time of 6 months)
Overall Survival | Following the last treatment, patient's condition will be monitored every 3 months until death.

CONTACTS AND LOCATIONS:
Overall Officials: Saul Rivkin, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (5):
- United States (5):
  - Swedish Cancer Institute Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute Issaquah Campus, Issaquah, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center Cancer Institute, Seattle, Washington
  - Swedish Cancer Institute Ballard Campus, Seattle, Washington

REFERENCES:
- [Derived] Rivkin SE, Moon J, Iriarte DS, Bailey E, Sloan HL, Goodman GE, BonDurant AE, Velijovich D, Wahl T, Jiang P, Shah CA, Drescher C, Fer MF, Kaplan HG, Ellis ED. Phase Ib with expansion study of olaparib plus weekly (Metronomic) carboplatin and paclitaxel in relapsed ovarian cancer patients. Int J Gynecol Cancer. 2019 Feb;29(2):325-333. doi: 10.1136/ijgc-2018-000035. Epub 2019 Jan 29. PMID 30700568